CLINICAL TRIAL: NCT01428284
Title: An Open-Label, Fixed-Sequence Study to Assess the Effects of Multiple-Dose Probenecid on the Multiple-Dose Pharmacokinetics of Canagliflozin in Healthy Subjects
Brief Title: A Study to Assess the Effects of Multiple-Dose Probenecid on the Multiple-Dose Pharmacokinetics of Canagliflozin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Director, Clinical Pharmacology, Johnson & Johnson Pharmaceutical Research and Development, L.L.C
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR018736; 28431754DIA1048 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C)
Record Dates: First submitted 2011-09-01; First posted 2011-09-02 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: Healthy Volunteers; Canagliflozin (JNJ-28431754); Pharmacokinetic; Probenecid
MeSH Terms: interventions — Canagliflozin; Probenecid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental): Canagliflozin/Probenecid
  Interventions: Drug: Canagliflozin/Probenecid

INTERVENTIONS:
Drug: Canagliflozin/Probenecid — Canagliflozin: Type = 1, unit = mg, number = 300, form = tablet, route = oral use. Probenicid: Type = 1, unit = mg, number = 500, form = tablet, route = oral use. One 300-mg canagliflozin tablet taken orally once daily on Days 1 to 14 (administration of canagliflozin alone) and on Days 15 to 17 (administration of canagliflozin + twice-daily administration of probenecid).

SUMMARY:
The purpose of this study is to assess the effects of multiple doses of probenecid on the multiple-dose pharmacokinetics of canagliflozin and its metabolites in healthy volunteers. Safety and tolerability will also be assessed.

DETAILED DESCRIPTION:
This will be a single-center, open-label (identity of study treatments will be known to volunteers participating in the study as well as to study staff) study to assess the effects of multiple doses of probenecid on the multiple-dose pharmacokinetics of canagliflozin and its metabolites in healthy volunteers. The study will last up to approximately 49 days (includes a Screening Phase of up to 19 days, an Open-Label Treatment Phase of 20 days, and a Post-Treatment Phase of up to 7 to 10 days). Healthy volunteers will take orally (by mouth) one 300 mg canagliflozin tablet once daily and/or one 500-mg probenecid tablet twice daily in sequential order as follows: Days 1 to 14 (administration of canagliflozin alone) and Days 15 to 17 (administration of canagliflozin + twice-daily administration of probenecid). On days when both canagliflozin and probenecid are taken, both doses must be taken at approximately the same time.

ELIGIBILITY:
Inclusion Criteria: Body mass index (BMI) between 18 and 28 kg/m² inclusive and a body weight of not less than 50 kg. Exclusion Criteria:History of or current medical illness, abnormal values for hematology or clinical chemistry laboratory tests, or abnormal physical examination, vital signs or 12-lead electrocardiogram (ECG) deemed to be clinically significant by the Investigator

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of Canagliflozin (including canagliflozin metabolites) | Up to Day 18
Plasma concentrations of probenecid | Up to Day 17

SECONDARY OUTCOMES:
Adverse Events | Up to 10 days following Day 18
  The number and type of adverse events
Clinical Laboratory Tests | Up to 10 days following Day 18
  Clinically relevant changes occurring in laboratory safety parameters
Vital Signs | Up to 10 days following Day 18
  Blood pressure and pulse

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Overland Park, Kansas, United States